CLINICAL TRIAL: NCT00677781
Title: The Impact of Microparticles on Inflammatory Responses During Visceral and Cardiac Surgery
Brief Title: Impact of Microparticles on Postoperative Complications in Surgical Patients
Status: Completed | Type: Observational
Sponsor: University of Bern (Other)
Responsible Party: Guido Beldi, MD, Department of visceral and transplant surgery, Inselspital Bern, Switzerland
Other Study IDs: KEK251_07
Record Dates: First submitted 2008-05-08; First posted 2008-05-15 (Estimated); Last update posted 2011-09-07 (Estimated); Status verified 2011-09

CONDITIONS: Neoplasm, Hepatic; Pancreatic Neoplasms; Colorectal Neoplasms
MeSH Terms: conditions — Liver Neoplasms; Pancreatic Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- F64: We investigate a cohort of 20 consecutive patients undergoing hepatic or pancreatic surgery (Pilot study)

SUMMARY:
Microparticles are cellular fragments which are released actively or passively under conditions of inflammation and stress. The impact of surgical operations on quantity and quality of microparticles remains unknown. In this observatory study we investigate quantitative and qualitative aspects of microparticles during cardiac and abdominal operations.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing cardiac or abdominal operations with a minimum expected operative time of 2 hours

Exclusion Criteria:

* Laparoscopic operations
* emergency operations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing cardiac or hepatobiliary or colorectal surgery. Setting: university hospital.
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2008-02; Primary Completion 2008-12 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Postoperative morbidity | 30 days

SECONDARY OUTCOMES:
Hospital stay | 30 days
Mortality | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Guido Beldi, MD, Principal Investigator — Bern University Hospital
Locations (1):
- Department of visceral and transplant surgery, Bern University Hospital, Bern, Switzerland

REFERENCES:
- [Background] Diamant M, Tushuizen ME, Sturk A, Nieuwland R. Cellular microparticles: new players in the field of vascular disease? Eur J Clin Invest. 2004 Jun;34(6):392-401. doi: 10.1111/j.1365-2362.2004.01355.x. PMID 15200490
- [Background] Piccin A, Murphy WG, Smith OP. Circulating microparticles: pathophysiology and clinical implications. Blood Rev. 2007 May;21(3):157-71. doi: 10.1016/j.blre.2006.09.001. Epub 2006 Nov 22. PMID 17118501
- [Background] Fujimi S, Ogura H, Tanaka H, Koh T, Hosotsubo H, Nakamori Y, Kuwagata Y, Shimazu T, Sugimoto H. Activated polymorphonuclear leukocytes enhance production of leukocyte microparticles with increased adhesion molecules in patients with sepsis. J Trauma. 2002 Mar;52(3):443-8. doi: 10.1097/00005373-200203000-00005. PMID 11901317
- [Background] Nieuwland R, Berckmans RJ, McGregor S, Boing AN, Romijn FP, Westendorp RG, Hack CE, Sturk A. Cellular origin and procoagulant properties of microparticles in meningococcal sepsis. Blood. 2000 Feb 1;95(3):930-5. PMID 10648405
- [Background] Ogura H, Kawasaki T, Tanaka H, Koh T, Tanaka R, Ozeki Y, Hosotsubo H, Kuwagata Y, Shimazu T, Sugimoto H. Activated platelets enhance microparticle formation and platelet-leukocyte interaction in severe trauma and sepsis. J Trauma. 2001 May;50(5):801-9. doi: 10.1097/00005373-200105000-00005. PMID 11371835
- [Background] Soriano AO, Jy W, Chirinos JA, Valdivia MA, Velasquez HS, Jimenez JJ, Horstman LL, Kett DH, Schein RM, Ahn YS. Levels of endothelial and platelet microparticles and their interactions with leukocytes negatively correlate with organ dysfunction and predict mortality in severe sepsis. Crit Care Med. 2005 Nov;33(11):2540-6. doi: 10.1097/01.ccm.0000186414.86162.03. PMID 16276178
- [Background] Boulanger CM, Scoazec A, Ebrahimian T, Henry P, Mathieu E, Tedgui A, Mallat Z. Circulating microparticles from patients with myocardial infarction cause endothelial dysfunction. Circulation. 2001 Nov 27;104(22):2649-52. doi: 10.1161/hc4701.100516. PMID 11723013
- [Background] Heloire F, Weill B, Weber S, Batteux F. Aggregates of endothelial microparticles and platelets circulate in peripheral blood. Variations during stable coronary disease and acute myocardial infarction. Thromb Res. 2003 Jun 1;110(4):173-80. doi: 10.1016/s0049-3848(03)00297-4. PMID 14512078
- [Background] Morel O, Hugel B, Jesel L, Lanza F, Douchet MP, Zupan M, Chauvin M, Cazenave JP, Freyssinet JM, Toti F. Sustained elevated amounts of circulating procoagulant membrane microparticles and soluble GPV after acute myocardial infarction in diabetes mellitus. Thromb Haemost. 2004 Feb;91(2):345-53. doi: 10.1160/TH03-05-0294. PMID 14961163
- [Background] Morel O, Jesel L, Freyssinet JM, Toti F. Elevated levels of procoagulant microparticles in a patient with myocardial infarction, antiphospholipid antibodies and multifocal cardiac thrombosis. Thromb J. 2005 Oct 11;3:15. doi: 10.1186/1477-9560-3-15. PMID 16219103
- [Background] van der Zee PM, Biro E, Ko Y, de Winter RJ, Hack CE, Sturk A, Nieuwland R. P-selectin- and CD63-exposing platelet microparticles reflect platelet activation in peripheral arterial disease and myocardial infarction. Clin Chem. 2006 Apr;52(4):657-64. doi: 10.1373/clinchem.2005.057414. Epub 2006 Jan 26. PMID 16439610
- [Background] Ardoin SP, Shanahan JC, Pisetsky DS. The role of microparticles in inflammation and thrombosis. Scand J Immunol. 2007 Aug-Sep;66(2-3):159-65. doi: 10.1111/j.1365-3083.2007.01984.x. PMID 17635793
- [Background] Andoh A, Tsujikawa T, Hata K, Araki Y, Kitoh K, Sasaki M, Yoshida T, Fujiyama Y. Elevated circulating platelet-derived microparticles in patients with active inflammatory bowel disease. Am J Gastroenterol. 2005 Sep;100(9):2042-8. doi: 10.1111/j.1572-0241.2005.50381.x. PMID 16128950
- [Background] Chamouard P, Desprez D, Hugel B, Kunzelmann C, Gidon-Jeangirard C, Lessard M, Baumann R, Freyssinet JM, Grunebaum L. Circulating cell-derived microparticles in Crohn's disease. Dig Dis Sci. 2005 Mar;50(3):574-80. doi: 10.1007/s10620-005-2477-0. PMID 15810645
- [Background] Jimenez JJ, Jy W, Mauro LM, Horstman LL, Soderland C, Ahn YS. Endothelial microparticles released in thrombotic thrombocytopenic purpura express von Willebrand factor and markers of endothelial activation. Br J Haematol. 2003 Dec;123(5):896-902. doi: 10.1046/j.1365-2141.2003.04716.x. PMID 14632781
- [Background] Proulle V, Hugel B, Guillet B, Grunebaum L, Lambert T, Freyssinet JM, Dreyfus M. Circulating microparticles are elevated in haemophiliacs and non-haemophilic individuals aged <18 years. Br J Haematol. 2005 Nov;131(4):487-9. doi: 10.1111/j.1365-2141.2005.05792.x. PMID 16281940